CLINICAL TRIAL: NCT03599557
Title: Improving HPV Vaccination Delivery in Pediatric Primary Care: The STOP-HPV Trial 1. Comparison of Communication Skills and Standard of Care for Uptake of the HPV Vaccine
Brief Title: The STOP-HPV Trial 1: Communication Intervention
Acronym: STOP-HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, Executive Vice-Chair and Vice-Chair for Research, Department of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01CA202261 (NIH); R01CA202261 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Immunization; Vaccination
Keywords: HPV; Vaccination; Practice based intervention

STUDY DESIGN:
Intervention Model Description: This study will use a cluster RCT study design to test the impact of the communication intervention to reduce missed opportunities (MOs) and raise HPV vaccine rates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Arm 1 will receive the STOP-HPV communication intervention
  Interventions: Behavioral: STOP-HPV communication intervention
- Control (No Intervention): Arm 2 will receive standard of care

INTERVENTIONS:
Behavioral: STOP-HPV communication intervention — This intervention will be communication skills training.
  Arms: Intervention

SUMMARY:
Most adolescents who receive human papillomavirus (HPV) vaccine are vaccinated in pediatric practices, yet missed opportunities (MOs) for HPV vaccination occur often and lead to low HPV vaccination rates. This cluster randomized clinical trial (RCT) will test the effectiveness (and cost-effectiveness) of training providers on HPV vaccine communication to reduce MOs and increase HPV vaccination rates.

DETAILED DESCRIPTION:
As highlighted by NCI, low HPV vaccination rates represent a major lost opportunity for population-wide cancer prevention. Pediatric primary care office visits are the main site for HPV vaccination, yet many missed opportunities (MOs) for vaccination occur in primary care and contribute to low vaccination rates. MOs are office visits during which a patient is eligible for a vaccine, but does not receive it. Many factors cause MOs - provider factors (e.g., time-constrained visits, lack of communication skills, and giving vaccinations only at preventive visits) and parent factors (e.g., vaccine hesitancy). This cluster randomized clinical trial will test the effectiveness (and cost-effectiveness) of training providers in HPV vaccine communication to reduce MOs and increase HPV vaccination rates. This training will be done through online educational modules (sent via text or email), weekly mini lessons and live office practice sessions.

ELIGIBILITY:
Practice Inclusion Criteria:

* The practice provides HPV vaccination services to adolescents.
* The practice is part of Physician's Computer Company (PCC), Office Practicum (OP) or (a) yet-to-be selected health system(s).
* The practice has had the same EHR system in place for a year or more (with special consideration on a case by case basis if they are close to but not do not reach a year).
* The practice agrees to not participate in other HPV-related QI projects or research interventions during the study period (with special consideration on a case by case basis).

Practice Exclusion Criteria:

* The practice plans to change EHR systems in the next three years.
* The practice participated in the last year, is currently engaged in, or plans to participate in an office-based HPV-related quality improvement (QI) project or research intervention during the study period (with special consideration on a case by case basis).
* Estimated 20% or more of adolescents at the practice receive HPV vaccinations at schools or health department clinics (given standard practice and published data, the investigators expect that few to no practices will need to be excluded based on this restriction).

Patient inclusion criteria:

-All patients of participating practices (intervention and comparison) aged 11-17 years who have at least 1 visit to the practice within the past two years.

Patient exclusion criteria:

-None apart from age of patients (above).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiks AG, Hannan C, Localio R, Kelly MK, Stephens-Shields AJ, Grundmeier RW, Shone LP, Steffes J, Breck A, Wright M, Rand CM, Albertin C, Humiston SG, McFarland G, Abney DE, Szilagyi PG. HPV Vaccinations at Acute Visits and Subsequent Adolescent Preventive Visits. Pediatrics. 2022 Nov 1;150(5):e2022058188. doi: 10.1542/peds.2022-058188. No abstract available. PMID 36205071
- [Derived] Szilagyi PG, Humiston SG, Stephens-Shields AJ, Localio R, Breck A, Kelly MK, Wright M, Grundmeier RW, Albertin C, Shone LP, Steffes J, Rand CM, Hannan C, Abney DE, McFarland G, Kominski GF, Seixas BV, Fiks AG. Effect of Training Pediatric Clinicians in Human Papillomavirus Communication Strategies on Human Papillomavirus Vaccination Rates: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2021 Sep 1;175(9):901-910. doi: 10.1001/jamapediatrics.2021.0766. PMID 34028494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Practices were recruited through the American Academy of Pediatrics' PROS (Pediatric Research in Office Settings) Network. Practices were the unit of randomization (48 practices total- 24 randomized into each arm).
Pre-assignment Details: The unit of randomization in this cluster randomized design is the practice. Eligible patients of the practices had at least one visit in the baseline and/or communication period in this cluster-randomized design (overlap between periods is possible).
Units Other Than Participants: Practices
Period: Baseline Period (12 Months)
Arm/Group | Intervention | Control
Started | 50569; 24 Practices | 53869; 24 Practices
Completed | 50569; 24 Practices | 53869; 24 Practices
Not Completed | 0; 0 Practices | 0; 0 Practices
Period: Communication Intervention (6 Months)
Arm/Group | Intervention | Control
Started | 29206; 24 Practices | 33914; 24 Practices
Completed | 29206; 24 Practices | 33914; 24 Practices
Not Completed | 0; 0 Practices | 0; 0 Practices

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants includes the number of individuals, but from 2 separate time periods- the Baseline Period (12 months) and the Communication Intervention Period (6 months). In this cluster-randomized design, participants could have had a visit in either or both periods.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 79775 | 87783 | 167558
Age, Customized [Count of Participants; unit: Participants]
  Adolescents ages 11-17 years: Baseline Period | 50569 | 53869 | 104438
  Adolescents ages 11-17 years: Communication Intervention | 29206 | 33914 | 63120
Sex/Gender, Customized [Count of Participants; unit: Participants] — The Overall Number of Baseline Participants includes the number of individuals, but from 2 separate time periods- the Baseline Period (12 months) and the Communication Intervention Period (6 months). In this cluster-randomized design, participants could have had one or more visits to their practice in either or both periods. Population: Participants in the baseline analysis population included the number of adolescents of the randomized practices who were aged 11-17 years with an eligible visit (HPV vaccine due), but from 2 separate time periods- the Baseline Period (12 mo) and Communication Intervention Period (6 mo). In this cluster-randomized design, participants could have had a visit in either or both periods. The sum of the two periods will equal the Overall Number of Baseline Participants provided above.
  Participants
    Baseline Period: number analyzed (Participants) | 50569 | 53869 | 104438
    Baseline Period: Male | 25472 | 27106 | 52578
    Baseline Period: Female | 25093 | 26762 | 51855
    Baseline Period: Missing | 4 | 1 | 5
    Communication Intervention: number analyzed (Participants) | 29206 | 33914 | 63120
    Communication Intervention: Male | 14542 | 16845 | 31387
    Communication Intervention: Female | 14664 | 17068 | 31732
    Communication Intervention: Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Overall Number of Baseline Participants includes the number of unique participants, but in 2 separate time periods- the Baseline Period (12 months) and the Communication Intervention Period (6 months). In this cluster-randomized design, participants could have had a visit in either or both periods.
  Participants
    Baseline Period: number analyzed (Participants) | 50569 | 53869 | 104438
    Baseline Period: White | 36054 | 31058 | 67112
    Baseline Period: African American | 4962 | 5080 | 10042
    Baseline Period: Asian or Pacific Islander | 2734 | 1901 | 4635
    Baseline Period: American Indiana/Alaskan Native | 229 | 448 | 677
    Baseline Period: Multiracial group | 348 | 352 | 700
    Baseline Period: Other | 178 | 223 | 401
    Baseline Period: Missing data | 6064 | 14807 | 20871
    Communication Intervention: number analyzed (Participants) | 29206 | 33914 | 63120
    Communication Intervention: White | 20824 | 19480 | 40304
    Communication Intervention: African American | 2705 | 3042 | 5747
    Communication Intervention: Asian or Pacific Islander | 1583 | 1148 | 2731
    Communication Intervention: American Indiana/Alaskan Native | 138 | 281 | 419
    Communication Intervention: Multiracial group | 215 | 223 | 438
    Communication Intervention: Other | 101 | 128 | 229
    Communication Intervention: Missing data | 3640 | 9612 | 13252

OUTCOME MEASURES:

1. Primary Outcome: Change in the Rate of Missed Vaccination Opportunities Among All Clinicians
Description: The difference in the missed opportunity rate for HPV vaccination between the baseline period (12 months long) and the feedback period (6 months long) among all the clinicians in the participating practices, regardless of whether they received the training intervention. A missed opportunity is a visit-based measure, with the denominator representing all the visits where an HPV vaccine is due at the time of the visit and the numerator representing the number of visits where an HPV vaccine was not given.
Time Frame: Assessment of rates from 2 time periods- baseline period (assessed outcomes retrospectively from minus 12 months to Time 0), followed by 6 month intervention period (excluding a 4 week ramp-up period).
Population: The Overall Number Participants analyzed is the number of unique patients with one or more visits to their practice (regardless of whether HPV vaccine was due) a study period - the Baseline Period (12 months) and the Communication Intervention Period (6 months). The number of units analyzed, serving as the denominator, is the number of eligible visits (visits where a child is due for HPV vaccine). The number of these visits where the vaccine was not given at the eligible visit is the numerator.
Measure: Count of Units; unit: Eligible visits (due for vaccine)
Units Other Than Participants: Eligible visits (due for vaccine)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 58279 | 62465
Number analyzed (Eligible visits (due for vaccine)) | 72372 | 80331
Eligible visits (due for vaccine)
  Baseline Period Missed Opportunity Rate: number analyzed (Participants) | 50569 | 53869
  Baseline Period Missed Opportunity Rate: number analyzed (Eligible visits (due for vaccine)) | 51339 | 55502
  Baseline Period Missed Opportunity Rate | 37063 | 40764
  Communication Intervention Missed Opportunity Rate: number analyzed (Participants) | 29206 | 33914
  Communication Intervention Missed Opportunity Rate: number analyzed (Eligible visits (due for vaccine)) | 21033 | 24829
  Communication Intervention Missed Opportunity Rate | 14932 | 18343

2. Primary Outcome: Change in the Rate of Missed Vaccination Opportunities Among Consenting Clinicians
Description: The difference in the missed opportunity rate for HPV vaccination between the baseline period (12 months long) and the feedback period (6 months long) among all the clinicians in the participating practices who received the training intervention. A missed opportunity is a visit-based measure, with the denominator representing all the visits where an HPV vaccine is due at the time of the visit and the numerator representing the number of visits where an HPV vaccine was not given.
Time Frame: as for outcome 1
Population: The unique children who made a visit (not just an HPV eligible visit) in either the baseline period (12 month) and/or the communication intervention period (6 month) to a clinician who consented to receive online training. Because the missed opportunity rate is a visit-based outcome, the overall number of units analyzed is the number of HPV eligible visits made in the two time periods and the count of units below is the number of visits where an HPV vaccination was not given in each period
Measure: Count of Units; unit: Eligible visits (HPV due)
Units Other Than Participants: Eligible visits (HPV due)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 46600 | 50585
Number analyzed (Eligible visits (HPV due)) | 50936 | 56598
Eligible visits (HPV due)
  Baseline Period: number analyzed (Eligible visits (HPV due)) | 35156 | 38508
  Baseline Period | 25117 | 27817
  Communication Intervention Period: number analyzed (Eligible visits (HPV due)) | 15780 | 18090
  Communication Intervention Period | 11152 | 13193

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected. This was not a drug/device trial, but a trial assessing the impact of provider education on missed opportunity rates.
Description: Adverse Events were not collected. This was not a drug/device trial, but a trial assessing the impact of provider education on missed opportunity rates.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03599557/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03599557/ICF_001.pdf